CLINICAL TRIAL: NCT04647162
Title: Safety of Surgical Treatment In Severe Primary Pontine Hemorrhage Evacuation (STIPE): a Multicentric, Randomized, Controlled, Open-label Trial
Brief Title: A Clinical Trial About the Safety of Surgical Treatment in Severe Primary Pontine Hemorrhage
Acronym: STIPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chao You, MD, former director of the department of neurosurgery, West China Hospital, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STIPE
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Cerebrovascular Disorders; Pontine Hemorrhage; Primary; Surgery
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: A sample size of 60 would be required to demonstrate a significant level of 5% (two-sided) with 80% power. Considering the 6% missing rate during follow-up, the total sample size was 64 cases with 16 and 48 cases in MT and HE group, respectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medical group (Active Comparator): Patients receive only medical treatment including active life support, nutritional support, homeostasis maintenance of the internal environment, and other symptomatic treatment.
  Interventions: Other: life support
- surgical group (Experimental): Patients receive intervention such as the evacuation of hematoma under craniotomy or by stereotactic puncture or neuroendoscopy.
  Interventions: Procedure: hematoma evacuation by craniotomy; Procedure: hematoma evacuation by stereotactic puncture; Procedure: hematoma evacuation by neuroendoscopy

INTERVENTIONS:
Procedure: hematoma evacuation by craniotomy — The intervention method of hematoma evacuation is under craniotomy.
  Arms: surgical group
Procedure: hematoma evacuation by stereotactic puncture — The intervention method of hematoma evacuation is under stereotactic puncture.
  Arms: surgical group
Procedure: hematoma evacuation by neuroendoscopy — The intervention method of hematoma evacuation is under neuroendoscopy.
  Arms: surgical group
Other: life support — The treatments in medical group includes life support, nutrition support, and rehabilitation therapy。
  Arms: medical group

SUMMARY:
Primary pontine hemorrhage (PPH) is not common but is the most catastrophic subtype of intracerebral hemorrhage, with acute mortality between 30% and 60%. For severe PPH, defined as Glasgow Coma score (GCS) <8 and hematoma volume≥5ml, the mortality rate is as high as 80-100%. Guidelines from the American Heart Association and European Stroke Organization do not make definite specifications. More than a century after Finkelnburg first explored the brainstem for hematoma, however, plenty of researches have shown surgery can save lives and improve the prognosis for selective patients and can be an effective and safe treatment. This study is proposed to validate the safety of surgical treatment in severe primary pontine hemorrhage.

DETAILED DESCRIPTION:
The study is being conducted from Jan 2022 to Nov 2024 in 20 neurosurgical units. This STIPE trial is an investigator-initiated, parallel (3:1 to surgical HE or MT), multi-centre, randomized controlled open-label trial following the Consolidated Standards of Reporting Trials (CONSORT) guidelines and will be conducted from Jan 2022 to Nov 2024 in 20 Tertiary hospitals in China. The flow chart of the clinical trial is presented in Figure 1. Neurosurgeons involved in the study are senior investigators with good clinical experience in sPPH management. Moreover, all investigators are well trained centrally according to the requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PPH: patients have acute hemorrhage mainly in pons with a definite history of hypertension.
2. GCS 5~7 and HV≥5ml on admission (the HV in intraventricular system being excluded).
3. Family members consenting to randomize and signing informed consent form (ICF).
4. Time from onset to admission less than 24 hours.
5. Age:18 years or older.

Exclusion Criteria:

1. Structural lesions such as brainstem cavernous malformation, arteriovenous malformation, aneurysm, tumor apoplexy.
2. GCS≥8 and HV<5ml.
3. Time from onset to admission over 24 hours.
4. Patients with platelet count < 100,000, International Normalized Ratio (INR)> 1.4, or an elevated prothrombin time (PT) and activated partial thromboplastin time (APTT).
5. Multiple ICH.
6. Accompanying hydrocephalus that requires surgical management
7. Irreversible brainstem failure (bilateral fixed, dilated pupils and extensor motor posturing, GCS≤4).
8. A previous history of ICH.
9. Any serious concurrent illness that would interfere with the safety assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease.
10. Pregnant patients.
11. Patients' family members refuse HE.
12. Any other condition that the investigator believes would present a significant hazard to the subject if the investigational therapy were initiated.
13. Participating in another simultaneous trial of ICH treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on the identity card
Enrollment: 64 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome Number 1: Rate of Mortality | 30 days from randomization
  Percentage of participants who died during the first 30 days after randomization.
Safety Outcome Number 2: Rate of Cerebritis, Meningitis, Bacterial Ventriculitis | 30 days from randomization
  Percentage of participants who had a bacterial brain infection (cerebritis, meningitis, ventriculitis) within 30 days of randomization.
Safety Outcome Number 3: Rate of Symptomatic Rebleeding | 72 hours post surgery
  The difference in the rate of symptomatic rebleeding 72 hours post surgery.

SECONDARY OUTCOMES:
the rate of hematoma clearance 3 days after surgery | 3 days after surgery
  the rate of hematoma clearance 3 days after surgery
all-cause mortality at 365 days | 365 days after surgery
  all-cause mortality at 365 days
neurological functional status of 30 days, 90 days, 180 days, and 365 days measured by Modified Rankin Scale (mRS), GCS and GOS. | 30 days, 90 days, 180 days, and 365 days after surgery
  neurological functional status of 30 days, 90 days, 180 days, and 365 days measured by Modified Rankin Scale (mRS), GCS and GOS.
The Extended Glasgow Outcome Scale (EGOS) at 180 days and 365 days | 180 days and 365 days after surgery
  The Extended Glasgow Outcome Scale (EGOS) at 180 days and 365 days
The 5-level EuroQol five dimensions questionnaire (EQ-5D) version (EQ-5D-5L) at 180 days and 365 days | 180 days and 365 days after surgery
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The former descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The latter is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.
the National Institutes of Health Stroke Scale (NIHSS) at 180 days and 365 days | 180 days and 365 days after surgery
  the National Institutes of Health Stroke Scale (NIHSS) at 180 days and 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Chao You, MD, Principal Investigator — West China Hospital
Locations (20):
- China (20):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Gaozhou Hospital of Traditional Chinese Medicine Affiliated to Guangzhou University of Chinese Medicine, Gaozhou, Guangdong
  - Guangdong Sanjiu Brain Hospital, Guangzhou, Guangdong
  - University of Chinese Academy of Sciences Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of South China University of Technology, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - General Hospital of the Eastern Theater, Nanjing, Jiangsu
  - Shanxi Bethune hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - The Third Hospital of the People's Liberation Army, Baoji
  - The seventh medical center of the Army General Hospital, Beijing
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Huashan Hospital of Fudan University, Shanghai
  - Shanghai No.10 hospital, Shanghai
  - Xuhui Hospital of Zhongshan Hospital affiliated to Fudan, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morotti A, Jessel MJ, Brouwers HB, Falcone GJ, Schwab K, Ayres AM, Vashkevich A, Anderson CD, Viswanathan A, Greenberg SM, Gurol ME, Romero JM, Rosand J, Goldstein JN. CT Angiography Spot Sign, Hematoma Expansion, and Outcome in Primary Pontine Intracerebral Hemorrhage. Neurocrit Care. 2016 Aug;25(1):79-85. doi: 10.1007/s12028-016-0241-2. PMID 26759226
- [Background] Ye Z, Huang X, Han Z, Shao B, Cheng J, Wang Z, Zhang Z, Xiao M. Three-year prognosis of first-ever primary pontine hemorrhage in a hospital-based registry. J Clin Neurosci. 2015 Jul;22(7):1133-8. doi: 10.1016/j.jocn.2014.12.024. Epub 2015 May 14. PMID 25982189
- [Background] Tao C, Li H, Wang J, You C. Predictors of Surgical Results in Patients with Primary Pontine Hemorrhage. Turk Neurosurg. 2016;26(1):77-83. doi: 10.5137/1019-5149.JTN.12634-14.1. PMID 26768872
- [Background] Huang K, Ji Z, Sun L, Gao X, Lin S, Liu T, Xie S, Zhang Q, Xian W, Zhou S, Gu Y, Wu Y, Wang S, Lin Z, Pan S. Development and Validation of a Grading Scale for Primary Pontine Hemorrhage. Stroke. 2017 Jan;48(1):63-69. doi: 10.1161/STROKEAHA.116.015326. Epub 2016 Dec 8. PMID 27932606
- [Background] Indredavik B, Bakke F, Slordahl SA, Rokseth R, Haheim LL. Stroke unit treatment. 10-year follow-up. Stroke. 1999 Aug;30(8):1524-7. doi: 10.1161/01.str.30.8.1524. PMID 10436094
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Steiner T, Al-Shahi Salman R, Beer R, Christensen H, Cordonnier C, Csiba L, Forsting M, Harnof S, Klijn CJ, Krieger D, Mendelow AD, Molina C, Montaner J, Overgaard K, Petersson J, Roine RO, Schmutzhard E, Schwerdtfeger K, Stapf C, Tatlisumak T, Thomas BM, Toni D, Unterberg A, Wagner M; European Stroke Organisation. European Stroke Organisation (ESO) guidelines for the management of spontaneous intracerebral hemorrhage. Int J Stroke. 2014 Oct;9(7):840-55. doi: 10.1111/ijs.12309. Epub 2014 Aug 24. PMID 25156220
- [Background] Lui TN, Fairholm DJ, Shu TF, Chang CN, Lee ST, Chen HR. Surgical treatment of spontaneous cerebellar hemorrhage. Surg Neurol. 1985 Jun;23(6):555-8. doi: 10.1016/0090-3019(85)90002-3. PMID 3992454
- [Background] Ichimura S, Bertalanffy H, Nakaya M, Mochizuki Y, Moriwaki G, Sakamoto R, Fukuchi M, Fujii K. Surgical Treatment for Primary Brainstem Hemorrhage to Improve Postoperative Functional Outcomes. World Neurosurg. 2018 Dec;120:e1289-e1294. doi: 10.1016/j.wneu.2018.09.055. Epub 2018 Sep 19. PMID 30244074
- [Background] Mangiardi JR, Epstein FJ. Brainstem haematomas: review of the literature and presentation of five new cases. J Neurol Neurosurg Psychiatry. 1988 Jul;51(7):966-76. doi: 10.1136/jnnp.51.7.966. PMID 3060565
- [Background] Rohde V, Berns E, Rohde I, Gilsbach JM, Ryang YM. Experiences in the management of brainstem hematomas. Neurosurg Rev. 2007 Jul;30(3):219-23; discussion 223-4. doi: 10.1007/s10143-007-0081-9. Epub 2007 May 8. PMID 17486379
- [Background] Murata Y, Yamaguchi S, Kajikawa H, Yamamura K, Sumioka S, Nakamura S. Relationship between the clinical manifestations, computed tomographic findings and the outcome in 80 patients with primary pontine hemorrhage. J Neurol Sci. 1999 Aug 15;167(2):107-11. doi: 10.1016/s0022-510x(99)00150-1. PMID 10521548
- [Background] Cao S, Zheng M, Hua Y, Chen G, Keep RF, Xi G. Hematoma Changes During Clot Resolution After Experimental Intracerebral Hemorrhage. Stroke. 2016 Jun;47(6):1626-31. doi: 10.1161/STROKEAHA.116.013146. Epub 2016 Apr 28. PMID 27125525
- [Background] Wilkinson DA, Keep RF, Hua Y, Xi G. Hematoma clearance as a therapeutic target in intracerebral hemorrhage: From macro to micro. J Cereb Blood Flow Metab. 2018 Apr;38(4):741-745. doi: 10.1177/0271678X17753590. Epub 2018 Jan 19. PMID 29350086
- [Background] Parraga RG, Possatti LL, Alves RV, Ribas GC, Ture U, de Oliveira E. Microsurgical anatomy and internal architecture of the brainstem in 3D images: surgical considerations. J Neurosurg. 2016 May;124(5):1377-95. doi: 10.3171/2015.4.JNS132778. Epub 2015 Oct 30. PMID 26517774
- [Derived] He Q, Wang J, Ma L, Li H, Tao C, You C. Safety of surgical Treatment In severe primary Pontine haemorrhage Evacuation (STIPE): study protocol for a multi-centre, randomised, controlled, open-label trial. BMJ Open. 2022 Aug 23;12(8):e062233. doi: 10.1136/bmjopen-2022-062233. PMID 35998952